CLINICAL TRIAL: NCT02487121
Title: Improving Weight Loss Maintenance Through Alternative Schedules of Treatment
Acronym: ImWeL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Associate Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23DK081607 (NIH)
Record Dates: First submitted 2015-06-26; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- variable interval schedule (Experimental): 12 group-based extended care treatment sessions scheduled in 3, 4-week periods over a 12-month period
  Interventions: Behavioral: variable interval schedule
- self-directed treatment (Active Comparator): provision of treatment materials with instruction to work through materials at participant's own pace
  Interventions: Behavioral: self-directed treatment

INTERVENTIONS:
Behavioral: variable interval schedule — 12 group-based extended care treatment sessions scheduled in 3, 4-week periods over a 12-month period
  Arms: variable interval schedule
Behavioral: self-directed treatment — provision of treatment materials with instruction to work through materials at participant's own pace
  Arms: self-directed treatment

SUMMARY:
This project examines the effects of differing schedules of extended care contact following weight loss treatment in order to prevent weight regain following treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years-old
* body mass index (BMI) = 28.0 - 45.0 kg/m2
* willing to provide informed consent and accept randomization

Exclusion Criteria:

* BMI >45 kg/m2
* Illnesses requiring medical attention and/or conditions for which weight loss and moderate physical activity would be inadvisable: diabetes not under active treatment, myocardial infarction or cerebrovascular accident within the last six months; unstable angina within the past six months; congestive heart failure; cancer requiring treatment in past five years (exception: non-melanoma skin cancer); serious infectious diseases (e.g., self-reported HIV); chronic hepatitis; cirrhosis; chronic malabsorption syndrome; chronic pancreatitis; chronic lung diseases that limit physical activity; orthopedic injuries or conditions that significantly limit physical activity.
* Conditions or behaviors likely to affect the conduct of the trial: unwilling or unable to give informed consent; unable to read English at the 5th grade level; unwilling to accept random assignment; unwilling or unable to travel to attend intervention (due to distance from clinic, work schedule or other scheduling conflicts); likely to relocate out of the service area in next 18 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
body weight (kg) | 12 months
  change in body weight (kg) between randomization and month-12 follow-up

REFERENCES:
- [Derived] Schneider-Worthington CR, Kinsey AW, Tan F, Zhang S, Borgatti AC, Davis AL, Dutton GR. Pretreatment and During-Treatment Weight Trajectories in Black and White Women. Am J Prev Med. 2022 Jul;63(1 Suppl 1):S67-S74. doi: 10.1016/j.amepre.2022.01.031. PMID 35725143
- [Derived] Dutton GR, Gowey MA, Tan F, Zhou D, Ard J, Perri MG, Lewis CE. Comparison of an alternative schedule of extended care contacts to a self-directed control: a randomized trial of weight loss maintenance. Int J Behav Nutr Phys Act. 2017 Aug 15;14(1):107. doi: 10.1186/s12966-017-0564-1. PMID 28806992